CLINICAL TRIAL: NCT05295303
Title: Quality Improvements in Post-Myocardial Infarction Management Using Home-Based RemOte Monitoring System (QIBO)
Brief Title: Home-based Remote Monitoring
Acronym: QIBO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung-Wah David SIU, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QIBO_1
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: To assess efficacy of home-based remote monitoring in post-myocardial infarction patient for improving guideline directed treatment utility, compared between subjects with home-based remote monitoring and management care (Interventional group) and conventional care (Control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Subjects will be provided with a home-based remote integrated post-MI management system and will be instructed to perform daily routine measurements. Site investigators will review the physiological parameters of patients randomized to the Intervention group daily and treatment can be initiated or modified accordingly through instant communication (electronic communication and/or phone).
  Interventions: Device: Remote integrated post-MI management system
- Control group (Placebo Comparator): Subjects will be provided with a home-based remote integrated post-MI management system and will be instructed to perform daily routine measurements. Site investigators will review individual patient physiological parameters and risk factors only during the clinic visits
  Interventions: Device: Remote integrated post-MI management system

INTERVENTIONS:
Device: Remote integrated post-MI management system — The home-based remote integrated post-MI management system comprises (1) a patch-based long-term Holter monitoring system HC3A250 (BISA Technologies (Hong Kong) Limited, Hong Kong SAR, China), (2) a handheld single-lead electrocardiogram (ECG) recorder (Comfit Healthcare Devices Limited, Hong Kong SAR, China), (3) a blood pressure monitor, (4) a patient-facing smartphone application specially designed for the study, and (5) a web-based clinical management system for clinicians
  Other Names: Holter monitoring system HC3A250 (BISA Technologies (Hong Kong) Limited, Hong Kong SAR, China); Single-lead electrocardiogram (ECG) recorder (Comfit Healthcare Devices Limited, Hong Kong SAR, China)

SUMMARY:
Acute myocardial infarction (MI) is a disease of high morbidity and mortality. It is usually caused by atherothrombosis of major epicardial coronary arteries which result in myocardial necrosis. Due to improvement in care systems, availability of revascularizations and better medical treatment, the mortality of MI has generally declined in the past 20 years. Nevertheless, patients survived MI are still at heightened risk of further cardiovascular events and death. Therefore, guideline directed secondary preventive measures are of paramount importance to improve long term outcome. These include adherence to medications and dose titration, risk factor modification, detection of arrhythmia and use of implantable cardio-defibrillator (ICD) as appropriate. In reality, guideline adherence is unsatisfactory and may lead to worse clinical outcomes. The underlying reasons are multi-factorial, including lack of patient education, recognition, motivation or physician inertia. Therefore, newer initiatives are required to reinforce secondary preventive measures.

In current era of health information technology, remote monitoring and telecommunication emerge to be practice-changing in various aspects of healthcare provision. Particularly for post MI survivors, the early post discharge period is vulnerable and a significant number of patients are readmitted 30 days after leaving hospital. This is not surprising as patients are still in recovering phase on medications titration and many of them may not fully accept they are suffering from a life-threatening condition. Besides, malignant arrhythmia may develop without the protection of ICD which is usually implanted after 40 days post MI as per clinical guidelines. As such, home-based remote monitoring with handheld single-lead electrocardiogram and patch-based continuous holter monitor can potentially detect arrhythmia which prompt early clinical attention. Furthermore, daily blood pressure measurement using dedicated smartphone applications enables physicians and patients to up-titrate medications to desired doses more quickly. This can hopefully strengthen compliance to better achieve guideline recommended treatment targets.

In the Quality Improvements in Post-Myocardial Infarction Management using Home-Based RemOte Monitoring System trial (QIBO; "岐伯" in Chinese), we investigate the feasibility and efficacy of utilizing a home-based remote monitoring system in post MI survivors. We hypothesize that this approach is effective to improve guideline directed treatment utility, cardiovascular risk factors target achievement and clinical outcome.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-labelled, randomized controlled trial. Patients with acute myocardial infarction with primary or early percutaneous coronary intervention (PCI) will be recruited upon hospital discharge. Patients with ST-segment elevation myocardial infarction (STEMI) and non-STEMI will be randomized in a 1:1 ratio to home-based remote management care (Intervention group) or conventional care (Control group) for 17 weeks.

Upon hospital discharge, all patients will be provided with a home-based remote integrated post-MI management system and will be instructed to perform daily routine measurements. Patients randomized to the Intervention group will be given patch-based Holter ECG monitoring till post-MI day 40.

The home-based remote integrated post-MI management system comprises (1) a patch-based long-term Holter monitoring system, (2) a handheld single-lead electrocardiogram (ECG) recorder, (3) a blood pressure monitor, (4) a patient-facing smartphone application specially designed for the study, and (5) a web-based clinical management system for clinicians.

All remotely obtained Holter data will be transferred daily via the study smartphone application to detect (1) ventricular arrhythmia, (2) ST-segment change, and (3) atrial fibrillation. Thereafter patients in the Interventional group will be instructed to record a 30-second single-lead ECG using the handheld ECG device every morning or when symptomatic. Patients in both the Intervention group and Control group will be instructed to measure their blood pressure in the morning and evening and input the data through the study smartphone application. All remotely obtained physiological data will be automatically transmitted in real-time to a secured cloud hosting and displayed on a web-based dashboard at the clinicians' offices. Physiological parameters of patients in the Interventional group will be reviewed daily by site investigators with preset algorithms to titrate or modify guideline directed medical therapy through instant communication (electronic communication and/or phone), whereas for the Control group, patient data will be reviewed only at the clinic visits. All patients will be followed up for 17 weeks.

There will have instruction session for study participants, a study research nurse will educate them on individual cardiovascular risk factors, life-style modification, and the treatment targets. In addition, the risk of recurrent cardiovascular event will be estimated using the Thrombolysis In Myocardial Infarction (TIMI) Risk Score for Secondary Prevention (TRS 2°P) score. The TRS 2°P incorporates 9 readily available clinical characteristics: congestive heart failure, hypertension, diabetes mellitus, age ≥75 years, prior stroke, prior coronary artery bypass graft, peripheral artery disease, estimated glomerular filtration rate <60, and smoking to predict recurrent cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized with acute myocardial infarction as defined as a detection of a rise and/or fall of troponin with at least 1 value above the 99th percentile upper reference limit together with either (1) symptoms of myocardial ischemia, or (2) ECG changes compatible with myocardial ischemia
* Treated with PCI for culprit lesson
* Voluntarily agrees to participate by providing written informed consent

Exclusion Criteria:

* Complex congenital heart disease
* Significant valvular stenosis
* Left ventricular assist device
* Listed for heart transplant
* Renal impairment with serum creatinine ≥ 190 μmol/L or on renal replacement therapy
* Inability or refusal to provide inform consent
* Short life expectance (< 1 year) due to concomitant medical condition(s)
* Lack of skills in operating simple electronic devices
* Unavailability of a mobile network service in the place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Renin-angiotensin-aldosterone system blockers | 17 weeks
  Percentage of patients with ≥50% maximal targeted dose (MTD) of renin-angiotensin-aldosterone system blockers

SECONDARY OUTCOMES:
Beta-adrenergic blockers | 17 weeks
  Percentage of patients with ≥50% maximal targeted dose (MTD) of beta-adrenergic blocker2
Ivabradine | 17 weeks
  Percentage of patients with ≥50% maximal targeted dose (MTD) of ivabradine
Statin | 17 weeks
  Percentage of patients with ≥50% maximal targeted dose (MTD) of statin
Renin-angiotensin-aldosterone system blockers | 17 weeks
  Dosage in terms of percentage maximal targeted dose (MTD) of renin-angiotensin-aldosterone system blockers
Beta-adrenergic blockers | 17 weeks
  Dosage in terms of percentage maximal targeted dose (MTD) of beta-adrenergic blockers
Ivabradine | 17 weeks
  Dosage in terms of percentage maximal targeted dose (MTD) of ivabradine
Statin | 17 weeks
  Dosage in terms of percentage maximal targeted dose (MTD) of statin
Low density lipoprotein | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of low density lipoprotein (< 1.4 mmol/L or >50% reduction)
High density lipoprotein | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of high density lipoprotein (> 1.0 mmol/L)
Triglyceride | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of triglyceride (< 1.7 mmol/L)
Body mass index | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of body mass index (< 25 kg/m2)
Resting blood pressure | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of resting blood pressure (systolic blood pressure within 100 - 120 mmHg and diastolic blood pressure within 60 - 90 mmHg)
Resting heart rate | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of resting heart rate (sinus rhythm 50 - 70 bpm and atrial fibrillation 50 - 110 bpm)
Hemoglobin A1C | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of hemoglobin A1c (< 7%)
Smoking cessation | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of smoking cessation
Moderate intensity aerobic exercise | 17 weeks
  Occurrence of achieving cardiovascular risk factors target of moderate intensity aerobic exercise (> equivalent of 30 minutes for 5 times per week)
Major adverse cardiovascular events | 17 weeks
  Occurrence of cardiovascular events of composite major adverse cardiovascular events including cardiovascular death from any causes, non-fatal myocardial infarction, unplanned coronary revascularization, and non-fatal stroke
Heart failure hospitalization | 17 weeks
  Occurrence of cardiovascular events of heart failure hospitalization
New-onset atrial fibrillation | 17 weeks
  Occurrence of cardiovascular events of new-onset atrial fibrillation
Sudden cardiac arrest | 17 weeks
  Occurrence of cardiovascular events of sudden cardiac arrest
Implantation of automatic implantable cardioverter-defibrillator | 17 weeks
  Occurrence of cardiovascular events of implantation of automatic implantable cardioverter-defibrillator
All cause mortality | 17 weeks
  Occurrence of cardiovascular events of all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Wah David Siu, Prof, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided